CLINICAL TRIAL: NCT02483364
Title: A Phase II Clinical Trial to Assess the Effect of HC-SVT-1001 (Autologous Fat Stem Adult Mesenchymal Cells Expanded and Combined With a Tricalcium Phosphate Biomaterial) and HC-SVT-1002 (Allogeneic Fat Stem Adult Mesenchymal Cells Expanded and Combined With a Tricalcium Phosphate Biomaterial) in the Surgical Treatment of Atrophic Pseudarthrosis of Long Bones
Brief Title: A Clinical Trial to Assess the Effect of HC-SVT-1001 and HC-SVT-1002 in the Surgical Treatment of Atrophic Pseudarthrosis of Long Bones (Bonecure)
Acronym: Bonecure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Salvat (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STEMQUIRI/12ES01
Record Dates: First submitted 2015-04-15; First posted 2015-06-26 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Pseudoarthrosis
MeSH Terms: conditions — Pseudarthrosis | interventions — Clinical Protocols

STUDY DESIGN:
Intervention Model Description: Cell therapy
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental (Experimental): HC-SVT-1001. Intraosseous use. 3x10(6) cells/cm3. (Initial protocol) HC-SVT-1002. Intraosseous use. 3x10(6) cells/cm3. (Protocol amendment)
  Interventions: Other: HC-SVT-1001(initial protocol); HC-SVT-1002 (protocol amendment)

INTERVENTIONS:
Other: HC-SVT-1001(initial protocol); HC-SVT-1002 (protocol amendment) — A single application in the context of a single surgical intervention.

SUMMARY:
The purpose os this study is to evaluate the safety and effectiveness of HC-SVT-1001 and HC-SVT-1002 in the surgical treatment of atrophic nonunion in long bones.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either sex between 18 and 65 years of age (both inclusive).
* Diagnosis of atrophic pseudoarthrosis of long bones confirmed radiographically.

Exclusion Criteria:

* Present infection (infection signs should not be evidenced).
* Other lesions which interfere with the body weight load.
* Open pseudoarthrosis (at the time of inclusion).
* Congenital bone diseases (hypophosphatemia), metabolic bone disease associated with primary or secondary hypoparathyroidism.
* Other conditions or circumstances that compromise the study participation according to medical criteria.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-11-10 (Actual); Primary Completion 2020-05-18 (Actual); Study Completion 2020-10-20 (Actual)

PRIMARY OUTCOMES:
Safety of HC-SVT-1001 and HC-SVT-1002 in the surgical treatment of atrophic nonunion in long bones by recording of adverse events. | Up to 24 months after surgery.
Effectiveness by mean of radiological methods on the appearance of signs of osseous setting formation. | Within 6 months after surgery.

SECONDARY OUTCOMES:
Comparative statistical analysis | Up to 24 months after surgery.
  Comparative statistical analysis between the 12 patients of this study and the data of 14 consecutive cases of refractory nonunion of long bones that have been treated since Sept-2009 with 40x10(6) autologous fat stem adult mesenchymal and under AEMPS compassionate use requirements.

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Jimenez, MD, Study Chair — Laboratorios Salvat
Locations (1):
- Laboratorios Salvat, S.A., Esplugues de Llobregat, Barcelone, Spain

REFERENCES:
- [Derived] Orozco Delclos L, Soler Rich R, Arriaza Loureda R, Moreno Garcia A, Gomez Barrena E. Efficacy and safety of autologous or allogeneic mesenchymal stromal cells from adult adipose tissue expanded and combined with tricalcium phosphate biomaterial for the surgical treatment of atrophic nonunion of long bones: a phase II clinical trial. J Transl Med. 2024 May 24;22(1):493. doi: 10.1186/s12967-024-05280-x. PMID 38789992